CLINICAL TRIAL: NCT03581708
Title: Real-world Study of the Incidence and Risk Factors of Venous Thromboembolism (VTE) in Chinese Advanced Stage Lung Cancer
Brief Title: Venous Thromboembolism in Advanced Lung Cancer
Acronym: RIVAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: No.GDREC 2018009H
Record Dates: First submitted 2018-05-25; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-05

CONDITIONS: Lung Neoplasms; Venous Thromboembolism
Keywords: lung cancer; Venous Thromboembolism
MeSH Terms: conditions — Lung Neoplasms; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 4 ml of peripheral blood is drawn from each subject and mononuclear cells are separated for DNA extraction, and mutation of Factor V Leiden will be examined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- advanced lung cancer: Patients diagnosed with advanced lung cancer
  Interventions: Other: lung cancer

INTERVENTIONS:
Other: lung cancer — If the patient is diagnosed with lung cancer in advanced stage, he/she will be followed up for VTE incidence
  Other Names: advance lung cancer

SUMMARY:
This is a prospective observatory clinical study, aiming to establish and validate venous thromboembolism risk model in Chinese advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
VTE has high incidence in lung cancer and increases the mortality. Appropriate preventive measures contribute to 50% increase of incidence. The investigators are to investigate the VTE in advanced non-small cell lung cancer and delineate the risk factors to establish a VTE risk model system helping clinicians to differentiate VTE high risk population and apply early prevention in order to reduce the incidence of VTE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of screening.
* Eastern Cooperative Oncology Group performance status of ≤ 2.
* Written informed consent obtained from the patient.
* Histologically and cytologically documented Stage 3B-4 lung cancer (according to Version 8 of the International Association for the Study of Lung Cancer Staging system).
* Patients with stage 1 to 3, who undergo radical therapy with disease free survival (DFS) >12 months.
* Willingness and ability to comply with scheduled visits and other study procedures.

Exclusion Criteria:

* History of another primary malignancy except for malignancy treated with curative intent with known active disease ≥ 5 years before date of the informed consent.
* Without signed informed consent.
* Unwillingness or inability to comply with scheduled visits or other study procedures.
* Previously diagnosed with VTE before signing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with advanced staged lung cancer with written informed consent.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
VTE incidence risk evaluation | 12 months
  Real world VTE incidence risk evaluation in advanced lung cancer. Establish and validate VTE risk predictive model in Chinese advanced lung cancer.

SECONDARY OUTCOMES:
VTE incidence | 12 months
  VTE incidence in advanced lung cancer.
VTE and overall survival | 12 months
  The influence on overall survival by VTE.

CONTACTS AND LOCATIONS:
Overall Officials: ZHEN WANG, Principal Investigator — Guangdong General Hospital, Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong General Hospital, Guangzhou, Guagndong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khorana AA, Kuderer NM, Culakova E, Lyman GH, Francis CW. Development and validation of a predictive model for chemotherapy-associated thrombosis. Blood. 2008 May 15;111(10):4902-7. doi: 10.1182/blood-2007-10-116327. Epub 2008 Jan 23. PMID 18216292
- [Result] Blom JW, Doggen CJ, Osanto S, Rosendaal FR. Malignancies, prothrombotic mutations, and the risk of venous thrombosis. JAMA. 2005 Feb 9;293(6):715-22. doi: 10.1001/jama.293.6.715. PMID 15701913
- [Result] Tesselaar ME, Osanto S. Risk of venous thromboembolism in lung cancer. Curr Opin Pulm Med. 2007 Sep;13(5):362-7. doi: 10.1097/MCP.0b013e328209413c. PMID 17940477
- [Result] Levitan N, Dowlati A, Remick SC, Tahsildar HI, Sivinski LD, Beyth R, Rimm AA. Rates of initial and recurrent thromboembolic disease among patients with malignancy versus those without malignancy. Risk analysis using Medicare claims data. Medicine (Baltimore). 1999 Sep;78(5):285-91. doi: 10.1097/00005792-199909000-00001. PMID 10499070
- [Result] Thodiyil PA, Kakkar AK. Variation in relative risk of venous thromboembolism in different cancers. Thromb Haemost. 2002 Jun;87(6):1076-7. No abstract available. PMID 12083490
- [Result] Stein PD, Beemath A, Meyers FA, Skaf E, Sanchez J, Olson RE. Incidence of venous thromboembolism in patients hospitalized with cancer. Am J Med. 2006 Jan;119(1):60-8. doi: 10.1016/j.amjmed.2005.06.058. PMID 16431186
- [Result] Chew HK, Davies AM, Wun T, Harvey D, Zhou H, White RH. The incidence of venous thromboembolism among patients with primary lung cancer. J Thromb Haemost. 2008 Apr;6(4):601-8. doi: 10.1111/j.1538-7836.2008.02908.x. Epub 2008 Jan 17. PMID 18208538
- [Result] Wang Z, Yan HH, Yang JJ, Wang BC, Chen HJ, Zhou Q, Xu CR, Jiang BY, Wu YL. Venous thromboembolism risk factors in Chinese non-small cell lung cancer patients. Support Care Cancer. 2015 Mar;23(3):635-41. doi: 10.1007/s00520-014-2405-y. Epub 2014 Aug 27. PMID 25155313